CLINICAL TRIAL: NCT07011966
Title: Evaluation of Adaptive Servo Ventilation Therapy for Insomnia Treatment Among Patients With Primary Insomnia
Brief Title: ASV Therapy for Insomnia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLP-25-01-01
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Insomnia; Insomnia (Moderate)
Keywords: Insomnia; ASV; PAP
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- ASV Therapy (Experimental)
  Interventions: Device: ASV therapy

INTERVENTIONS:
Device: ASV therapy — Adaptive servo ventilation (ASV) therapy using ResMed AirCurve 11 device will be used to target potential upper airway resistance and respiratory related arousals in patients with insomnia. The ASV device is approved for the treatment of obstructive sleep apnea, and this will be designated as the investigational device for this study with appropriate labelling.

SUMMARY:
This will be a single center, prospective study designed to evaluate the effect of adaptive servo ventilation therapy on insomnia severity among patients with moderate to severe chronic insomnia.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the effectiveness of adaptive servo ventilation therapy to reduce insomnia severity in primary insomnia patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Complaint of insomnia when presenting at clinic
* Diagnosis of moderate to severe insomnia through the Insomnia Severity Index (ISI) with a score ≥ 15
* Meet diagnostic criteria of Insomnia Disorder (per American Academy of Sleep Medicine)
* Naïve to treatment for sleep-disordered breathing (SDB), including CPAP, APAP, ASV; mandibular repositioning devices (MRDs), and any other nasal or oral therapy with a primary indication of treating SDB
* Owns a smartphone and is able to install an application for HSAT data syncing.
* Able to fully understand study information in English and sign informed consent

Exclusion Criteria:

* Primary complaint of sleep-disordered breathing or issues with apneas during sleep or excessive daytime sleepiness
* Pregnant or planning to be pregnant
* Any prior diagnosis of severe respiratory disorder or severe sleep disorder such as restless leg syndrome (RLS), idiopathic hypersomnia, or narcolepsy
* High risk for moderate to severe OSA based on STOP-BANG score.
* BMI > 40 kg/m2
* Anticipated changes to start or stop sedative or psychotropic medications during the course of the trial.
* Medical history of congestive heart failure (CHF) or other potentially unstable cardiac disease as well as chronic lung diseases or other debilitating medical conditions that manifest as more prominent in the patient's health compared to their sleep complaints.
* Daily use of opiate medications
* Known contraindications to PAP therapy as listed in the indication for use (i.e. heart failure (NYHA 2-4) with reduced left ventricular ejection fraction (LVEF ≤45%) and moderate to severe predominant central sleep apnea).
* Inability to pre-emptively comply with study procedures
* Patients who wish to continue using sleeping pills/hypnotics during the study
* Patients with conditions affecting the rotation of the condyle in the temporo-mandibular joint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) score | 4 weeks after therapy start
  Change in insomnia severity from baseline to 4 weeks after treatment initiation, as measured by subjective questionnaire

SECONDARY OUTCOMES:
Sleep Onset Latency | 4 weeks after treatment initiation
  Change in from baseline to end of treatment in sleep onset time

CONTACTS AND LOCATIONS:
Locations (1):
- C.S. Mott Center, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided